CLINICAL TRIAL: NCT05155657
Title: A Pilot Clinical Study to Evaluate Safety, Tolerability and Preliminary Efficacy of Intravenous Infusion of Umbilical Cord Mesenchymal Stem Cell in the Treatment of Decompensated Alcoholic Cirrhosis
Brief Title: Study of Decompensated Alcoholic Cirrhosis Treatment by Stem Cells
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yantai Yuhuangding Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-001
Record Dates: First submitted 2021-11-19; First posted 2021-12-13 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Alcoholic Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis, Alcoholic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low dose umbilical cord mesenchymal stem cells (UCMSCs) (Experimental)
  Interventions: Biological: Conventional therapy plus low dose UCMSCs treatment
- Medium dose UCMSCs (Experimental)
  Interventions: Biological: Conventional therapy plus medium dose UCMSCs treatment
- High dose UCMSCs (Experimental)
  Interventions: Biological: Conventional therapy plus high dose UCMSCs treatment

INTERVENTIONS:
Biological: Conventional therapy plus low dose UCMSCs treatment — Patients will receive the conventional therapy plus low dose UCMSCs treatment (0.5×10^6 UCMSCs/kg body)
  Arms: Low dose umbilical cord mesenchymal stem cells (UCMSCs)
Biological: Conventional therapy plus medium dose UCMSCs treatment — Patients will receive conventional therapy plus medium dose UCMSCs treatment (1×10^6 UCMSCs/kg body)
  Arms: Medium dose UCMSCs
Biological: Conventional therapy plus high dose UCMSCs treatment — Patients will receive conventional therapy plus high dose UCMSCs treatment (2×10^6 UCMSCs/kg body)
  Arms: High dose UCMSCs

SUMMARY:
The main purpose of this study is to evaluate the safety and tolerance of umbilical cord mesenchymal stem cells (UCMSCs) in patients with decompensated alcoholic cirrhosis, and to provide dose basis for subsequent clinical study design. We will also explore the possible mechanism of UCMSCs in the treatment of decompensated alcoholic cirrhosis (DAC).

DETAILED DESCRIPTION:
This study adopted a single-center, single-arm, single-dose combined multiple-dose administration, and dose-escalation clinical trial design to evaluate the safety, tolerability and preliminary effectiveness of UCMSCs in the treatment of patients with decompensated liver cirrhosis. Patients were recruited into three different dose groups, and 12 subjects were enrolled in each group. The subjects of each group will receive 0.5×10^6 cells/kg, 1.0×10^6 cells/kg, and 2.0×10^6 cells/kg respectively. According to the principle of dose escalation, subjects preset to low-dose will receive the administration first. Each group will receive only one corresponding dose for safety and tolerability check. The subjects will be observed for 21 days after the initial dose due to limited proliferation or differentiation potential and relatively low immunogenicity of mesenchymal stem cell products. The safety measures will be discussed by the Data Safety and Monitoring Board (DSMB) to determine whether subjects who have received a single dose will proceed with subsequent injections. Once all subjects in the lower-dose group have completed the initial administration and observed for 21 days. The DSMB will decided whether to proceed with the next-dose group. All subjects will receive routine drug treatment during the study. Primary endpoint: incidence and severity of cell therapy related adverse events from the beginning of treatment to the end of the follow-up. Secondary end point of the study includes: the change in Model For End-Stage Liver Disease (MELD) score of the subjects from baseline, at 1, 3, 6 and 12 months after the last administration; the overall survival rate at the 12th month after the last administration; Changes in liver function compared with baseline at 1, 3, 6 and 12 months after the last administration; changes of child Pugh score compared with baseline at 1, 3, 6 and 12 months after the last administration; and the change of Karnofsky Performance Status Scale (KPS) score from baseline at 1, 3, 6 and 12 months after the last administration.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18~60 years old;
2. The subject was diagnosed as decompensated alcoholic liver cirrhosis, according to the Guidelines for the Diagnosis and Treatment of Liver Cirrhosis and the Guidelines for the Prevention and Treatment of Alcoholic Liver Disease (2018);
3. The subject was previously diagnosed but treatment is ineffective;
4. Liver function was in child Pugh grade A or MELD score < 12;
5. Intermittent albumin supplementation and diuretic treatment are required;
6. The subject's Albumin level is less than 35g/L, total bilirubin is smaller than 10 times of the upper limit of normal value (hepatocyte hepatitis), or smaller than 15 times of the upper limit of normal value (cholestatic hepatitis or hepatocyte combined with cholestatic hepatitis), prothrombin activity is over 40% (grade II or lower hepatic encephalopathy has been controlled);
7. No history of gastrointestinal hemorrhage in the past month;
8. The subject understand and voluntarily sign the informed consent.

Exclusion Criteria:

1. The subject is allergic physique, with a history of drug or food allergies, especially those who are allergic to umbilical cord mesenchymal stem cells and any components in excipients;
2. The subject suffer acute attack of gastrointestinal bleeding, hepatic encephalopathy, hepatorenal syndrome or infection;
3. The subject suffer systemic infection or severe infection during screening;
4. Abnormal laboratory examinations results, including blood routine: peripheral blood white blood cell count <2.0×10^9/L or >12×10^9/L, hemoglobin (Hb) is less than 70% lower limit of the normal value, platelets <50×10^9/L ; Liver function: ALT or AST> 5 times the upper limit of normal; Renal function: Serum Creatinine (sCr)> 1.5 times the upper limit of normal; in case of abnormality, test shall be repeated;
5. Those who were positive for Hepatitis B surface Antigen (HBsAg) or Hepatitis C virus (HCV) antibody, Human Immunodeficiency Virus (HIV) antibody or syphilis antibody during screening;
6. Subjects suffer from serious, progressive, or uncontrolled diseases of important organs (including cardiovascular system, liver, lung and kidney), and other autoimmune diseases, malignant tumors, or a history of previous tumors, as well as other diseases that researchers believe that they are not suitable to participate in this clinical study.
7. Subject who has received stem cell therapy within 6 months before the screening;
8. Subject who has received biotherapy or participated in other clinical studies within 3 months before screening;
9. Female subjects who are pregnant, lactating, or premenopausal subject who failed to take medically approved non-drug contraceptive measures (such as intrauterine device, condom, female sterilization) during treatment and within 6 months after the treatment; or have a pregnancy plan within 6 months after the end of the study;
10. Male subjects who fail to take medically approved non-drug contraceptive measures (such as male sterilization or condom) during the treatment period and within 6 months after the end of the treatment;
11. Other factors that the researchers believe are not suitable for entering the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-06-13 (Actual); Primary Completion 2024-12-25 (Estimated); Study Completion 2024-12-25 (Estimated)

PRIMARY OUTCOMES:
Severity and incidence of adverse events (SIAE) on the 3rd day after the first administration | The 3rd day after the first administration
  According to the evaluation criteria of common adverse events (CTCAE v5.0), any AE occurred in all subjects during the clinical study, including abnormalities in clinical symptoms and vital signs and abnormalities in laboratory examination was observed.
1 week SIAE after the first administration | 1 week after the first administration
  According to the evaluation criteria of common adverse events (CTCAE v5.0), any AE occurred in all subjects during the clinical study, including abnormalities in clinical symptoms and vital signs and abnormalities in laboratory examination was observed.
3 weeks SIAE after the first administration | 3 week after the first administration
  According to the evaluation criteria of common adverse events (CTCAE v5.0), any AE occurred in all subjects during the clinical study, including abnormalities in clinical symptoms and vital signs and abnormalities in laboratory examination was observed.
3 week SIAE after the the second administration | 3 weeks after the the second administration
  According to the evaluation criteria of common adverse events (CTCAE v5.0), any AE occurred in all subjects during the clinical study, including abnormalities in clinical symptoms and vital signs and abnormalities in laboratory examination was observed.
1 month SIAE after the last administration | 1 month after the last administration
  According to the evaluation criteria of common adverse events (CTCAE v5.0), any AE occurred in all subjects during the clinical study, including abnormalities in clinical symptoms and vital signs and abnormalities in laboratory examination was observed.
3 months SIAE after the last administration | 3 months after the last administration
  According to the evaluation criteria of common adverse events (CTCAE v5.0), any AE occurred in all subjects during the clinical study, including abnormalities in clinical symptoms and vital signs and abnormalities in laboratory examination was observed.
6 months SIAE after the last administration | 6 months after the last administration
  According to the evaluation criteria of common adverse events (CTCAE v5.0), any AE occurred in all subjects during the clinical study, including abnormalities in clinical symptoms and vital signs and abnormalities in laboratory examination was observed.
12 months SIAE after the last administration | 12 months after the last administration
  According to the evaluation criteria of common adverse events (CTCAE v5.0), any AE occurred in all subjects during the clinical study, including abnormalities in clinical symptoms and vital signs and abnormalities in laboratory examination was observed.
24 months SIAE after the last administration | 24 months after the last administration
  According to the evaluation criteria of common adverse events (CTCAE v5.0), any AE occurred in all subjects during the clinical study, including abnormalities in clinical symptoms and vital signs and abnormalities in laboratory examination was observed.

SECONDARY OUTCOMES:
Child-Pugh score (effectiveness evaluation index) | At baseline, 3, 7 and 21 days after the first administration, 21 days after the second administration (if any), and 1, 3, 6 and 12 months after the last administration.
  The Child-Pugh grading standard is a grading standard commonly used in clinical practice to quantitatively evaluate the liver reserve function of patients with liver cirrhosis. Grading: 5~6 points for Grade A, 7~9 points for Grade B and 10~15 points for grade C;
  Note:
  For Primary Biliary Cirrhosis (PBC) or Primary Sclerosing Cholangitis (PSC): total bilirubin (umol/L): 17~68 is 1 point, 68~170 is 1 point, and >170 is 1 point; The Child-Pugh grading standard has been widely recognized by clinicians, and provides a specific clinical reference for the selection of treatment options for patients with liver cirrhosis and has important clinical value.
Survival rate (effectiveness evaluation index) | 12 months after the last administration.
  Overall survival rate of participants in this study.
Liver function (effectiveness evaluation index) | Baseline, 3, 7, and 21 days after the first administration, 21 days after the second administration (if any), and 1, 3, 6, and 12 months after the last administration.
  Indicators: Alanine transaminase (AST), Alanine transaminase (ALT)
The Model for End-Stage Liver Disease (MELD) score (effectiveness evaluation index) | Baseline, 3, 7, and 21 days after the first administration, 21 days after the second administration (if any), and 1, 3, 6, and 12 months after the last administration.
  MELD is a numerical scale, ranging from 6 (less ill) to 40 (gravely ill), used for liver transplant candidates age 12 and older. It gives each person a 'score' (number) based on how urgently he or she needs a liver transplant within the next three months.
  The number is calculated by a formula using three routine lab test results:
  MELD score = 3.8×ln[bilirubin (mg/dl)] + 11.2×ln(INR) + 9.6×ln[Scr(mg/dl)] + 6.4×(Cause: Bile or alcoholic 0, other 1) Bilirubin (mg/dl) = Bilirubin (μmol/L)/17.1 Scr(mg/dl) = Scr(μmol/L)/88.4
KPS score (effectiveness evaluation index) | Baseline, 3, 7, and 21 days after the first administration, 21 days after the second administration (if any), and 1, 3, 6, and 12 months after the last administration.
  KPS score is the Karnofsky (Karen, KPS, percentile method) functional status scoring standard. The higher the score, the better the health status, and the more the patient able to tolerate the side effects of treatment, hence a better curative effect. It is generally believed that a Karnofsky score above 80 is independent, which means the patient is able to take care of himself. Karnofsky score between 50 to 70 stands for a semi-independent status, that is, the patient is semi-self-care. A score of 50 means the patients require help from others. Those with a score greater than 80 are in better postoperative state and have a longer survival period.
  The lower the score, the worse the health status. If the score is less than 60, many effective anti-tumor treatments cannot be implemented.
Detection of Blood Coagulation Index of PT (effectiveness evaluation index) | Baseline, 3, 7, and 21 days after the first administration, 21 days after the second administration (if any), and 1, 3, 6, and 12 months after the last administration.
  To test the blood coagulation index of Prothrombin time (PT);
Detection of Blood Coagulation Index of APTT (effectiveness evaluation index) | Baseline, 3, 7, and 21 days after the first administration, 21 days after the second administration (if any), and 1, 3, 6, and 12 months after the last administration.
  To test the blood coagulation index of activated partial thromboplastin time (APTT);
Detection of Blood Coagulation Index of TT (effectiveness evaluation index) | Baseline, 3, 7, and 21 days after the first administration, 21 days after the second administration (if any), and 1, 3, 6, and 12 months after the last administration.
  To test the blood coagulation index of thrombin time (TT);
Detection of Blood Coagulation Index of FIB (effectiveness evaluation index) | Baseline, 3, 7, and 21 days after the first administration, 21 days after the second administration (if any), and 1, 3, 6, and 12 months after the last administration.
  To test the blood coagulation index of fibrinogen (FIB);

CONTACTS AND LOCATIONS:
Overall Officials: Jun Cui, MD, Principal Investigator — Yantai Yuhuangding Hospital
Locations (1):
- Yantai Yuhuangding Hospital, Yantai, Shandong, China